CLINICAL TRIAL: NCT07077681
Title: Acceptability and Therapeutic Maintenance of the Biosimilar Ustekinumab After Substitution
Brief Title: Evaluation of the Acceptability and Therapeutic Maintenance After Substitution of Ustekinumab With a Biosimilar
Status: Recruiting | Type: Observational
Sponsor: EG Labo (Industry)
Responsible Party: Sponsor
Other Study IDs: Etude ATLAS France 2025
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Crohn Disease (CD)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a population of adult patients followed for Crohn's disease, who had previously agreed to replace Stelara® with a biosimilar of ustekinumab (Uzpruvo®) and were followed over a period of 12 months under usual medical practice conditions.

* Main objective: To assess the maintenance of the biosimilar of ustekinumab at 12 months without returning to the reference treatment
* Secondary objectives:

  * To describe the factors associated with the maintenance of the biosimilar
  * To evaluate the evolution of patients' quality of life
  * To assess the rate of maintenance of clinical remission at M12
  * To describe the acceptability of the biosimilar treatment by patients
  * To evaluate patient satisfaction
  * To evaluate treatment tolerance
  * To describe the reasons for treatment discontinuation that occurred during follow-up
  * To describe the profile of patients who discontinued treatment upon their request.

DETAILED DESCRIPTION:
This is an open-label, prospective, longitudinal, multicenter, observational cohort study involving a population of adult patients for whom the investigating physician, prior to inclusion, decided with their consent to replace Stelara® with Uzpruvo® (a biosimilar of ustekinumab).

This observational study does not alter the physician-patient relationship or standard patient care. Physicians retain freedom in their prescriptions and follow-up procedures; no specific procedures or tests are required of patients beyond the completion of self-assessment questionnaires. The study is longitudinal, and the proposed assessments remain within the framework of the patients' standard follow-up with their physician.

This study is classified as RIPH 3 (minimally or not at all interventional).

The conduct of the treatment (dosage, administration schedule, etc.) is left to the discretion of the investigating physician in compliance with the MA, according to their clinical practice and the patient's therapeutic history. Similarly, the investigating physician remains the sole judge of the continuation or interruption of ustekinumab or its replacement by another biotherapy or by any other treatment. All treatments associated with ustekinumab as part of the management of the condition that prompted biotherapy that will be prescribed during the study must be reported in the observation log.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient who has agreed to participate in the study and does not oppose the use of their health data
* Patient with moderate to severe Crohn's disease treated with Stelara® in a pre-filled syringe according to the summary of product characteristics (SPC) with intervals of 8 or 12 weeks between injections
* Patients presenting at least one of the following objective criteria: o PCR < 5 mg/l o Calprotectin < 250 μg/g o Harvey-Bradshaw index < 5
* Patient in stable remission (defined by a stable ustekinumab dosage over the last 24 weeks and absence of corticosteroids for at least 3 months)• Patient for whom the investigator physician, prior to inclusion, has decided with their agreement, to replace Stelara® with Uzpruvo®
* Patient having internet access enabling them to complete online questionnaires

Exclusion Criteria:

* Patient treated with ustekinumab with intervals between injections less than 8 weeks
* Patients treated with ustekinumab in a pre-filled pen
* Patient included in an interventional clinical trial at the time of inclusion
* Patient refusing or unable to comply with the study follow-up procedures (patient unreachable by phone, unable to fill out the self-questionnaire or poorly speaking French...)
* Patient under legal protection, under guardianship or under curatorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Crohn disease treated by ustekinumab
Sampling Method: Non-Probability Sample
Enrollment: 246 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
maintenance of treatment | Month 12
  The maintenance of treatment is defined by the continuation of treatment with Uzpruvo®, the biosimilar of ustekinumab, during the twelve months of the study.

SECONDARY OUTCOMES:
Quality of life - SF-36 | Inclusion
  The Medical Outcomes Study Short-Form General Health Survey (SF-36) is a generic quality of life questionnaire. It consists of 36 questions concerning the four weeks preceding the survey, divided into eight dimensions: physical activity, life and relationships with others, physical pain, perceived health, vitality, limitations due to mental health, limitations due to physical health, and mental health.
Quality of life - SF-36 | Month 3
  The Medical Outcomes Study Short-Form General Health Survey (SF-36) is a generic quality of life questionnaire. It consists of 36 questions concerning the four weeks preceding the survey, divided into eight dimensions: physical activity, life and relationships with others, physical pain, perceived health, vitality, limitations due to mental health, limitations due to physical health, and mental health.
Quality of life - SF-36 | Month 6
  The Medical Outcomes Study Short-Form General Health Survey (SF-36) is a generic quality of life questionnaire. It consists of 36 questions concerning the four weeks preceding the survey, divided into eight dimensions: physical activity, life and relationships with others, physical pain, perceived health, vitality, limitations due to mental health, limitations due to physical health, and mental health.
Quality of life - SF-36 | Month 12
  The Medical Outcomes Study Short-Form General Health Survey (SF-36) is a generic quality of life questionnaire. It consists of 36 questions concerning the four weeks preceding the survey, divided into eight dimensions: physical activity, life and relationships with others, physical pain, perceived health, vitality, limitations due to mental health, limitations due to physical health, and mental health.
Quality of life - EQ-5D-5L | Inclusion
  The EQ-5D-5L questionnaire is a European quality of life scale comprising two parts: a first part with questions known as the "EQ-5D descriptive system," supplemented by a visual analog scale, called the "EQ-5D VAS." It consists of a 20 cm line, graduated from 0 to 100, on which the patient must indicate how they assess their current health, with 0 being the worst possible state and 100 the best.
Quality of life - EQ-5D-5L | Month 3
  The EQ-5D-5L questionnaire is a European quality of life scale comprising two parts: a first part with questions known as the "EQ-5D descriptive system," supplemented by a visual analog scale, called the "EQ-5D VAS." It consists of a 20 cm line, graduated from 0 to 100, on which the patient must indicate how they assess their current health, with 0 being the worst possible state and 100 the best.
Quality of life - EQ-5D-5L | Month 6
  The EQ-5D-5L questionnaire is a European quality of life scale comprising two parts: a first part with questions known as the "EQ-5D descriptive system," supplemented by a visual analog scale, called the "EQ-5D VAS." It consists of a 20 cm line, graduated from 0 to 100, on which the patient must indicate how they assess their current health, with 0 being the worst possible state and 100 the best.
Quality of life - EQ-5D-5L | Month 12
  The EQ-5D-5L questionnaire is a European quality of life scale comprising two parts: a first part with questions known as the "EQ-5D descriptive system," supplemented by a visual analog scale, called the "EQ-5D VAS." It consists of a 20 cm line, graduated from 0 to 100, on which the patient must indicate how they assess their current health, with 0 being the worst possible state and 100 the best.
Quality of life - SIBDQ | Inclusion
  The Short Inflammatory Bowel Disease Questionnaire is the abbreviated, self-administered version of the IBDQ, a quality of life questionnaire specific to IBD. It includes 10 questions exploring four domains: digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbances (3 items), and social function (2 items). As with the IBDQ, each item is assessed on a Likert scale. The total score ranges from 10 to 70. The higher the score, the better the quality of life.
Quality of life - SIBDQ | Month 3
  The Short Inflammatory Bowel Disease Questionnaire is the abbreviated, self-administered version of the IBDQ, a quality of life questionnaire specific to IBD. It includes 10 questions exploring four domains: digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbances (3 items), and social function (2 items). As with the IBDQ, each item is assessed on a Likert scale. The total score ranges from 10 to 70. The higher the score, the better the quality of life.
Quality of life - SIBDQ | Month 6
  The Short Inflammatory Bowel Disease Questionnaire is the abbreviated, self-administered version of the IBDQ, a quality of life questionnaire specific to IBD. It includes 10 questions exploring four domains: digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbances (3 items), and social function (2 items). As with the IBDQ, each item is assessed on a Likert scale. The total score ranges from 10 to 70. The higher the score, the better the quality of life.
Quality of life - SIBDQ | Month 12
  The Short Inflammatory Bowel Disease Questionnaire is the abbreviated, self-administered version of the IBDQ, a quality of life questionnaire specific to IBD. It includes 10 questions exploring four domains: digestive symptoms (3 items), systemic symptoms (2 items), emotional disturbances (3 items), and social function (2 items). As with the IBDQ, each item is assessed on a Likert scale. The total score ranges from 10 to 70. The higher the score, the better the quality of life.
Crohn's disease activity | Inclusion
  The Harvey-Bradshaw Index is the most widely used tool for assessing Crohn's disease activity in current practice. It comprises five items (general well-being, abdominal pain, number of loose stools per day, abdominal mass, and extradigestive signs). A score < 4 corresponds to inactive disease; a score between 4 and 12 to active disease; a score above 12 to very severe active disease.
Crohn's disease activity | Month 3
  The Harvey-Bradshaw Index is the most widely used tool for assessing Crohn's disease activity in current practice. It comprises five items (general well-being, abdominal pain, number of loose stools per day, abdominal mass, and extradigestive signs). A score < 4 corresponds to inactive disease; a score between 4 and 12 to active disease; a score above 12 to very severe active disease.
Crohn's disease activity | Month 6
  The Harvey-Bradshaw Index is the most widely used tool for assessing Crohn's disease activity in current practice. It comprises five items (general well-being, abdominal pain, number of loose stools per day, abdominal mass, and extradigestive signs). A score < 4 corresponds to inactive disease; a score between 4 and 12 to active disease; a score above 12 to very severe active disease.
Crohn's disease activity | Month 12
  The Harvey-Bradshaw Index is the most widely used tool for assessing Crohn's disease activity in current practice. It comprises five items (general well-being, abdominal pain, number of loose stools per day, abdominal mass, and extradigestive signs). A score < 4 corresponds to inactive disease; a score between 4 and 12 to active disease; a score above 12 to very severe active disease.
Abdominal pain | Inclusion
  The PRO-2 questionnaire consists of two separate questions (abdominal pain and stool frequency), each with four response options.
Abdominal pain | Month 3
  The PRO-2 questionnaire consists of two separate questions (abdominal pain and stool frequency), each with four response options.
Abdominal pain | Month 6
  The PRO-2 questionnaire consists of two separate questions (abdominal pain and stool frequency), each with four response options.
Abdominal pain | Month 12
  The PRO-2 questionnaire consists of two separate questions (abdominal pain and stool frequency), each with four response options.
Intestinal urgency | Inclusion
  The intestinal urgency questionnaire is an 11-point numeric self-assessment scale. The score increases with the severity of the urgency.
Intestinal urgency | Month 3
  The intestinal urgency questionnaire is an 11-point numeric self-assessment scale. The score increases with the severity of the urgency.
Intestinal urgency | Month 6
  The intestinal urgency questionnaire is an 11-point numeric self-assessment scale. The score increases with the severity of the urgency.
Intestinal urgency | Month 12
  The intestinal urgency questionnaire is an 11-point numeric self-assessment scale. The score increases with the severity of the urgency.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Cabinet Medical, Amiens
  - Chu de La Côte Basque, Bayonne
  - Chu Besançon - Hopital Jean Minjoz, Besançon
  - Chu La Cavale Blanche, Brest
  - Chu Montpellier - Hopital Saint Eloi, Montpellier
  - Chu Nantes, Nantes
  - Clinique Jules Verne, Nantes
  - Institut Des Mici Groupe Hospitalier, Neuilly-sur-Seine
  - Chu Lyon Sud, Pierre-Bénite
  - CHU Rouen Normandie, Rouen
  - Chu Nancy Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No